CLINICAL TRIAL: NCT03106454
Title: Ovulation Incidence in Oral Contraceptive Users
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Brian T. Nguyen, MD MSc, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HS-09-00669
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Contraception; Ovulation
MeSH Terms: interventions — Ethinyl Estradiol; Norethindrone Acetate; ferrous fumarate; norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination; Norethindrone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination oral contraceptive pill (Active Comparator): Ethinyl Estradiol 10mcg/Norethindrone acetate 1mg/ferrous fumarate 75mg Taken cyclically as 24 tablets containing EE 10mcg/NET acetate 1mg 2 tablets of EE 10mcg only 2 tablets of ferrous fumarate 75mg
  Interventions: Drug: Ethinyl Estradiol, Norethindrone acetate, ferrous fumarate
- Progestin only pill (Experimental): Norethindrone 0.35mg Marketed use for 1 tablet per day. For study dosing, patients will take 3 tablets daily for a total of 1.05mg daily.
  Interventions: Drug: Norethindrone

INTERVENTIONS:
Drug: Ethinyl Estradiol, Norethindrone acetate, ferrous fumarate — Combination Oral Contraceptive Pill. Ethinyl Estradiol 10mcg/Norethindrone acetate 1mg/ferrous fumarate 75mg
  Other Names: Loestrin
  Arms: Combination oral contraceptive pill
Drug: Norethindrone — Norethindrone 1.05mg
  Other Names: Micronor; Camilla
  Arms: Progestin only pill

SUMMARY:
Since the introduction of the combined hormonal contraceptive pill, dosages of ethinyl estradiol (EE) have steadily decreased from more than 150mcg to 20mcg in an attempt to improve the risk profile associated with the COC. In 2010, the Food and Drug Administration approved a oral contraceptive pill containing EE 10mcg/NET acetate 1mg (Tradename Lo loestrin). However, no studies have compared this formulation to pills containing either higher doses of estrogen or progestin alone. It is not known whether EE 10mcg is sufficient to prevent follicular development or to support the endometrium as well as higher doses of EE. This trial addresses the question of whether an oral contraceptive pill with EE 10mcg/Norethindrone acetate 1mg will better suppress ovulation or have a better side effect profile than a progestin only pill with a nearly equal dose of norethindrone.

DETAILED DESCRIPTION:
Use of combined hormonal contraceptives (CHC) containing estrogen is associated with venous thromboembolic events. In an effort to decrease the risks of estrogen, the dose of ethinyl estradiol (EE) contained in combined oral contraceptive (COC) pills has decrease substantially from >100mcg to 20mcg. In 2012, a COC with only 10mcg of EE (Tradename LoLoestrin) was approved by the Food and Drug Administration. However, no studies have compared this formulation to pills containing progestin alone to determine if this very low dose of EE decreases ovulation or improves unscheduled uterine bleeding beyond what is seen with a progestin only pill (POP).

We aim to compare a COC with EE 10mcg/norethindrone (NET) acetate 1mg to a POP containing a nearly equal amount of progestin (norethindrone 1.05mg). The objective of the study is to compare the incidence of ovulation among users of a COC with only EE10mcg/NET acetate 1mg to users of a POP with a nearly identical progestin dose of NET 1.05mg. We plan to recruit 58 women between the ages of 18 and 45 years old, who are ovulatory at baseline based on serum progesterone levels. Subjects will be randomized to take either a COC containing EE 10mcg/NET acetate 1mg or a POP containing NET 1.05mg for one month. During the month of study treatment, we will measure ovulation incidence using a single serum progesterone levels of >=4.0ng/dl, sperm penetration of cervical mucus using the Eggert Kruse classification system, pill compliance by NET serum levels, and side effects including unscheduled uterine bleeding via subject daily diaries.

Our primary outcome, ovulation incidence, will be compared between study arms. Secondary outcomes will compare cervical mucus quality, sperm penetration of cervical mucus, side effects (including uterine bleeding), and pill compliance between users of these two pills.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged women 18-45 years old.
* Menstrual cycle length 25-35days
* BMI less than or equal to 40
* English or Spanish speaking

Exclusion Criteria:

* Pregnant or breastfeeding in the previous 3 months.
* Use of OC, hormonal vaginal rings or patches, levonorgestrel containing intrauterine device, or etonogestrel implant in the previous 1 month. No use of depot medroxyprogesterone acetate (DMPA) injection in the previous 6 months and at least one menses since discontinuation.
* Medical contraindications to estrogen or progestin use. Specifically: smoking among participants over 35 years old, migraines with aura, history of blood clots, ischemic heart disease, stroke, breast cancer, cervical cancer, liver disease, symptomatic gallbladder disease, uncontrolled hypertension, antiphospholipid antibody syndrome, hyperlipidemia, diabetes with end organ damage (retinopathy, nephropathy, neuropathy) or diagnosis >20 years ago, organ transplant
* Desire to become pregnant in the next 4 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2024-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Ovulation | A single 28 day cycle
  Ovulation based on a single serum progesterone level of 4ng/dl or greater

SECONDARY OUTCOMES:
Sperm penetration of cervical mucus | A single 28 day cycle
  The average distance sperm will travel in vitro in a test tube of cervical mucus collected from the participant.
Cervical mucus quality | A single 28 day cycle
  Scoring of the ovulatory quality (thickness, cellularity, etc.) of cervical mucus collected from the participant
Side effects | A single 28 day cycle
  Side effects self reported by the participant
Uterine bleeding | A single 28 day cycle
  A daily calendar counting the number of days of uterine bleeding participants experience during the study cycle.

OTHER OUTCOMES:
Pill complaince | A single 28 day cycle
  Number of pills missed or forgotten over the course of a single 28 day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Nguyen, MD, MSc, Principal Investigator — University of Southern California
Locations (1):
- Brian T. Nguyen, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No